CLINICAL TRIAL: NCT00018304
Title: Insulin Action: Role of Skeletal Muscle and Insulin-Mediated Blood Flow
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: AGCG-005-98S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Hypertension
Keywords: blood pressure; insulin sensitivity; blood flow
MeSH Terms: conditions — Hypertension; Insulin Resistance

SUMMARY:
The overall objective of this proposal is to examine the contribution of changes in total body fat, enhancement in insulin-mediated vasodilatation and enhancement in endothelium-derived nitric oxide production to the improvements in metabolic insulin action. In addition, the study will track whether these improvements are related to changes in blood pressure.

ELIGIBILITY:
Age 50 - 75 years, elevated blood pressure, BMI greater than 25 but less than 40 kg/m2

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Leon, M.D.; Alan Blank, M.D.
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States